CLINICAL TRIAL: NCT02982668
Title: A Multi-center Randomised Controlled Trial to Explore the Ideal Initial Enteral Feeding Strategies in Patients With Severe Stroke at Acute Stage
Brief Title: Optimizing Early Enteral Nutrition in Severe Stroke
Acronym: OPENS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Significantly higher mortality
Sponsor: Xijing Hospital (Other)
Collaborators: Tang-Du Hospital (Other); Xi'an Central Hospital (Other); Xi'an Gaoxin Hospital (Other); Yan'an University Affiliated Hospital (Other); 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); Xi'an No.3 Hospital (Other Government); First Affiliated Hospital Xi'an Jiaotong University (Other); Yulin No.1 Hospital (Unknown); First People's Hospital of Xianyang (Other); Tongchuan Mining Hospital (Unknown); The PLA General Hospital of Xinjiang (Unknown); Tongchuan People's Hospital (Unknown); Yulin No.2 Hospital (Other); Ankang Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KY20162086-2
Record Dates: First submitted 2016-11-27; First posted 2016-12-05 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2020-12

CONDITIONS: Severe Stroke; Acute Stroke; Dysphagia
Keywords: severe stroke; Acute Stroke; Enteral Feeding; Mortality; Disability; Clinical trial
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Metoclopramide; mosapride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full enteral feeding (Active Comparator): The caloric goal of the first day is one-third of caloric requirements, the second day is half of caloric requirements, the third day is 70-100% and sustained for 1 week. Protein requirements are calculated at 1.2 to 1.5 g per kilogram of body weight per day.
  Interventions: Other: Initial enteral feeding
- Modified full enteral feeding (Experimental): Consistent with full enteral feeding plan, preventively add metoclopramide or mosapride everyday to improve gastrointestinal (GI) motility.
  Interventions: Other: Initial enteral feeding; Drug: metoclopramide or mosapride
- Permissive underfeeding (Experimental): The caloric goal of the first day is one-third of caloric requirements, the second day is 40-60% and sustained for 1 week. Protein requirements are calculated at 1.2 to 1.5 g per kilogram of body weight per day.
  Interventions: Other: Initial enteral feeding

INTERVENTIONS:
Other: Initial enteral feeding
Drug: metoclopramide or mosapride — gastrointestinal (GI) motility improving
  Arms: Modified full enteral feeding

SUMMARY:
The purpose of this academic lead study is to explore the ideal nutritional support strategy for patient with acute severe stroke.

DETAILED DESCRIPTION:
Of high mortality and morbidity, severe stroke is associated with devastating damages in neurologic, respiratory, circulatory and many other systems. The outcomes of patients with severe stroke depend largely on medical strategies on acute stage, especially on nutritional support management. Unfortunately, clinical evidence are sparse and the ideal initial feeding strategy remains disputable.

The IF-STROKE study aims to provide reliable data on the effects of modified full enteral feeding (target recruitment 200) and permissive underfeeding in patients with acute severe stroke (target recruitment 200) compared to full enteral feeding (target recruitment 200). Patients presenting with acute (<72h) severe stroke (GCS ≦ 12 or NIHSS ≧ 11) and dysphagia (defined by Water Swallowing Test) will be randomly assigned to full enteral feeding, modified full enteral feeding, or permissive underfeeding treatment for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Severe stroke occurred in 7 days.
* GCS ≤12 or NIHSS≥11.
* Any cases of profiles #3 through 5 in Water Swallowing Test or with disorder of consciousness.
* Plan to receive enteral feeding for at least 7 days.
* Informed consent.

Exclusion Criteria:

* Gastrointestinal diseases before stroke, such as gastrointestinal resection, malabsorption,and irritable bowel syndrome.
* Brain death.
* Complicated with the disease which only have life expectancy < 6 months in over 50% patients.
* After cardiac arrest.
* Received parenteral nutrition support.
* Pregnant woman.
* Concurrent severe hepatic or renal dysfunction。
* Unstable hemodynamics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Rate of patients with death or major disability (modified Rankin scale score ≥3) | 3 months after enrollment
  modified Rankin scale score, with score ranging from 0 (normal) to 6 (death), was used to evaluate the functional outcomes after stroke.

SECONDARY OUTCOMES:
Mortality (rate of patients with death) | 3 months after enrollment
  Rate of patients with death
The scores of National Institute of Health stroke scale | 7 days after enrollment
  National Institute of Health stroke scale, with scores ranging from 0 (normal function) to 42 (functional impairment)) was used to evaluate the impairment caused by a stroke.
Glasgow Coma Scale | 7 days after enrollment
  Glasgow Coma Scale, with scores ranging from 3 (no response) to 15 (normal response), was used to grade the conscious state.
modified Rankin scale | 7 days after enrollment
  modified Rankin scale score, with score ranging from 0 (normal) to 6 (death), was used to evaluate the functional outcomes after stroke.
Barthel index | 7 days after enrollment
  The Barthel Index is a scale, with score ranging from 0 to 100 (normal), that measures disability or dependence in activities of daily living in stroke patients
modified Rankin scale | 3 months after enrollment
  modified Rankin scale score, with score ranging from 0 (normal) to 6 (death), was used to evaluate the functional outcomes after stroke.
Barthel index | 3 months after enrollment
  The Barthel Index is a scale, with score ranging from 0 to 100 (normal), that measures disability or dependence in activities of daily living in stroke patients
The incidence of treatment intolerance | 7 days after enrollment
  The intolerance including gastric retention, diarrhea, constipation, gastrointestinal hemorrhage
The incidence of serious adverse events | 3 months after enrollment
The incidence of adverse events That are related to treatment | 3 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Wen Jiang, PhD, Study Director — Department of Neurology, Xijing Hospital, Fourth Military Medical University
Locations (4):
- China (4):
  - Xijing Hospital, Xi'an, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University,, Xi'an, Shaanxi
  - Yulin No.2 Hospital, Yunlin, Shaanxi

REFERENCES:
- [Background] Wirth R, Smoliner C, Jager M, Warnecke T, Leischker AH, Dziewas R; DGEM Steering Committee*. Guideline clinical nutrition in patients with stroke. Exp Transl Stroke Med. 2013 Dec 1;5(1):14. doi: 10.1186/2040-7378-5-14. PMID 24289189
- [Background] McClave SA, Taylor BE, Martindale RG, Warren MM, Johnson DR, Braunschweig C, McCarthy MS, Davanos E, Rice TW, Cresci GA, Gervasio JM, Sacks GS, Roberts PR, Compher C; Society of Critical Care Medicine; American Society for Parenteral and Enteral Nutrition. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Adult Critically Ill Patient: Society of Critical Care Medicine (SCCM) and American Society for Parenteral and Enteral Nutrition (A.S.P.E.N.). JPEN J Parenter Enteral Nutr. 2016 Feb;40(2):159-211. doi: 10.1177/0148607115621863. No abstract available. PMID 26773077
- [Result] FOOD Trial Collaboration. Poor nutritional status on admission predicts poor outcomes after stroke: observational data from the FOOD trial. Stroke. 2003 Jun;34(6):1450-6. doi: 10.1161/01.STR.0000074037.49197.8C. Epub 2003 May 15. PMID 12750536
- [Result] Ukleja A. Altered GI motility in critically Ill patients: current understanding of pathophysiology, clinical impact, and diagnostic approach. Nutr Clin Pract. 2010 Feb;25(1):16-25. doi: 10.1177/0884533609357568. PMID 20130154
- [Result] Dennis MS, Lewis SC, Warlow C; FOOD Trial Collaboration. Effect of timing and method of enteral tube feeding for dysphagic stroke patients (FOOD): a multicentre randomised controlled trial. Lancet. 2005 Feb 26-Mar 4;365(9461):764-72. doi: 10.1016/S0140-6736(05)17983-5. PMID 15733717
- [Result] Heyland DK, Stephens KE, Day AG, McClave SA. The success of enteral nutrition and ICU-acquired infections: a multicenter observational study. Clin Nutr. 2011 Apr;30(2):148-55. doi: 10.1016/j.clnu.2010.09.011. Epub 2010 Oct 25. PMID 20971534
- [Result] Jie B, Jiang ZM, Nolan MT, Zhu SN, Yu K, Kondrup J. Impact of preoperative nutritional support on clinical outcome in abdominal surgical patients at nutritional risk. Nutrition. 2012 Oct;28(10):1022-7. doi: 10.1016/j.nut.2012.01.017. Epub 2012 Jun 5. PMID 22673593
- [Result] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Rice TW, Wheeler AP, Thompson BT, Steingrub J, Hite RD, Moss M, Morris A, Dong N, Rock P. Initial trophic vs full enteral feeding in patients with acute lung injury: the EDEN randomized trial. JAMA. 2012 Feb 22;307(8):795-803. doi: 10.1001/jama.2012.137. Epub 2012 Feb 5. PMID 22307571
- [Result] Permissive Underfeeding or Standard Enteral Feeding in Critically Ill Adults. N Engl J Med. 2015 Sep 24;373(13):1281. doi: 10.1056/NEJMx150028. No abstract available. PMID 26398094
- [Derived] Sakai K, Niimi M, Momosaki R, Hoshino E, Yoneoka D, Nakayama E, Masuoka K, Maeda T, Takahashi N, Sakata N. Nutritional therapy for reducing disability and improving activities of daily living in people after stroke. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD014852. doi: 10.1002/14651858.CD014852.pub2. PMID 39145517
- [Derived] Zhao J, Yuan F, Song C, Yin R, Chang M, Zhang W, Zhang B, Yu L, Jia Y, Ma Y, Song Y, Wang C, Song C, Wang X, Shang L, Yang F, Jiang W; OPENS Trial Investigators. Safety and efficacy of three enteral feeding strategies in patients with severe stroke in China (OPENS): a multicentre, prospective, randomised, open-label, blinded-endpoint trial. Lancet Neurol. 2022 Apr;21(4):319-328. doi: 10.1016/S1474-4422(22)00010-2. Epub 2022 Feb 24. PMID 35219379
- [Derived] Yuan F, Yang F, Zhang W, Jia Y, Ma Y, Qu Y, Wang X, Huo K, Wang C, Yuan X, Song C, Zhang B, Jiang W; OPENS study group. Optimizing early enteral nutrition in severe stroke (OPENS): protocol for a multicentre randomized controlled trial. BMC Neurol. 2019 Feb 12;19(1):24. doi: 10.1186/s12883-019-1253-2. PMID 30755171